CLINICAL TRIAL: NCT02566291
Title: Supraglottic Airways LMA Supreme and Ambu AuraGain in Clinical Practice: a Prospective Observational Study
Brief Title: Observational Study With Investigation of Two Second Generation Laryngeal Masks
Acronym: OSSGA
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Marc Kriege, MD; Rüdiger Noppens, MD, Johannes Gutenberg University Mainz
Other Study IDs: SGA 2014
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Airway Remodeling
Keywords: laryngeal mask; airway leakage; airway morbidity
MeSH Terms: conditions — Airway Remodeling

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Supreme Group: Measuring Success rate and Insertion Time
  Interventions: Device: Success
- Gain Group: Measuring Success rate and Insertion Time
  Interventions: Device: Success

INTERVENTIONS:
Device: Success — Success rate and time for insertion

SUMMARY:
In a observational study the second-generation laryngeal masks LMA Supreme and Ambu AuraGain are investigated.

DETAILED DESCRIPTION:
After approval from the local ethics committee, data were collected in a prospective, non- randomised study over a three-month period. When contra-indications for laryngeal mask use were absent anaesthesiologists used either Supreme (Teleflex Medical GmbH, Germany) or Gain (Ambu GmbH, Germany). Endpoints were the success rate and time to insertion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years
* No concurrent participation in another study
* capacity to consent
* Present written informed consent of the research participant
* Elective surgery under general anesthesia

Exclusion Criteria:

* Age <18 years
* Existing pregnancy
* Lack of consent
* inability to consent
* emergency patients
* Emergency situations in the context of a Difficult Airway Management
* ASA classification> 3
* situations where the possibility of accumulated gastric contents
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  Age > 18 Years informed consent elective surgery undergoing general anesthesia non-pregnant
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2015-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Success rate | 70-98 Percent
  overall and first attempt success rate

SECONDARY OUTCOMES:
Time for insertion | 5-120 seconds
Leakage in ml.min | 0-300 ml.min

CONTACTS AND LOCATIONS:
Overall Officials: Marc MK Kriege, MD, Principal Investigator — University JG, Mainz
Locations (1):
- Department of Anaesthesiology;, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Russo SG, Cremer S, Galli T, Eich C, Brauer A, Crozier TA, Bauer M, Strack M. Randomized comparison of the i-gel, the LMA Supreme, and the Laryngeal Tube Suction-D using clinical and fibreoptic assessments in elective patients. BMC Anesthesiol. 2012 Aug 7;12:18. doi: 10.1186/1471-2253-12-18. PMID 22871204